CLINICAL TRIAL: NCT07015554
Title: Study on Serum IGF1 in Female Patients With Heart Failure With Preserved Ejection Fraction
Brief Title: Serum IGF1 on Female HFpEF Patients
Acronym: IGF1
Status: Enrolling by invitation | Type: Observational
Sponsor: The University of Hong Kong-Shenzhen Hospital (Other)
Responsible Party: Principal Investigator, Cai Sidong, Assistant Research Fellow, The University of Hong Kong-Shenzhen Hospital
Other Study IDs: 8230-1; 82300446 (Other Grant/Funding Number: National Science Foundation of China); RCBS20231211090745071 (Other Grant/Funding Number: Shenzhen Science and Technology Innovation Bureau)
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: HFpEF - Heart Failure With Preserved Ejection Fraction
Keywords: Insulin growth factor (IGF1); Heart failure with preserved ejection fraction (HFpEF)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study Title: Application of Serum IGF1 in the Diagnosis of Female Heart Failure with Preserved Ejection Fraction (HFpEF) Study Institution: Hong Kong University-Shenzhen Hospital Principal Investigator: Sidong Cai

1. Study Purpose This study aims to investigate whether serum insulin-like growth factor 1 (IGF1) can be used to improve the diagnosis of heart failure with preserved ejection fraction (HFpEF) in women, providing preliminary insights for early detection of this condition in female patients.
2. Study Procedures Information Collection: Relevant medical information will be collected during your outpatient visit or hospitalization.

   Subject Identification: If you agree to participate, you will be assigned a unique study number to establish a medical record file.

   Blood Sampling:

   Blood samples will be collected concurrently with routine clinical blood draws (no additional needle insertions).

   Volume: 10-20 mL of venous blood each time, collected on the enrollment day, 3 months, 6 months, and 12 months after enrollment.

   Use of Samples: Samples will be used exclusively for this study. Follow-up Examinations: Standard HF follow-up tests (e.g., echocardiograms) will be conducted as clinically necessary. These are part of routine HF management and will not impose extra burden on you.
3. Risks and Discomforts Confidentiality: All information will be kept strictly confidential.

   Minimal Risks:

   Temporary pain, bruising, or tenderness at the blood draw site. Rarely, mild dizziness or (extremely rarely) needle site infection.
4. Responsibilities as a Research Subject

   You are required to:

   Provide truthful information about your medical history and current health status. Report any discomfort experienced during the study to the research doctor. Avoid taking restricted medications or foods as instructed. Disclose if you are currently participating in, or have recently participated in, other research studies.
5. Privacy Protection Anonymization: Blood samples will be labeled with your study number, not your name.

   Confidentiality:

   Identifiable information will not be disclosed to anyone outside the research team without your permission. Research staff and the sponsor are obligated to maintain your privacy. Records will be stored in locked cabinets and accessible only to authorized researchers. Regulatory agencies or ethics committees may review your data (anonymized) to ensure study compliance. No personal identifying information will be disclosed in study publications.
6. Compensation for Study-Related Injuries In the event of a study-related injury, you are entitled to compensation in accordance with Chinese law.
7. Voluntary Participation and Withdrawal You may refuse to participate or withdraw from the study at any time. Withdrawal will not affect your medical care or rights. Data collected before withdrawal will be excluded from the study results upon your request.

   The researcher may terminate your participation if you fail to follow the protocol, require other treatments, experience study-related injuries, or for other medical reasons.
8. Contact Information For questions about the study, your rights, or any discomfort/injury during the study, please contact Principal Investigator: Dr. Sidong Cai via caisd@hku-szh.org.

ELIGIBILITY:
Inclusion Criteria:

* age over 18;
* female participants only;

Exclusion Criteria:

* with congenital heart disease or with other family disease history
* participants receiving hormone therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population was divided into two part: (1) Healthy population; (2) HFpEF population. For healthy population, candidates are female sex, age over 18, without any congenital heart defects or heart diseases. For HFpEF population, candidates are female sex, age over 18, with HFpEF diagnosis or all criteria mentioned below:
  * Clinical manifestations-Typical symptoms of heart failure (such as decreased activity tolerance, sitting breathing) or signs (such as moist rales in the lungs, edema of the lower extremities);
    * Left ventricular ejection fraction (LVEF) -LVEF ≥50% without significant dilation in the left ventricle;
      * Evidence of cardiac structural or functional abnormalities-LAVI>34 mL/m², LVMI >95 g/m², E/e' ratio >15, tricuspid regurgitation velocity >2.8 m/s, etc.
        * Biomarker: BNP≥35 pg/mL or NT-proBNP≥125 pg/mL (patients with sinus rhythm) ⑤ Without cardiac amyloidosis, hypertrophic cardiomyopathy, valvular heart disease, pericardial disease and lung/kidney disease
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
IGF1 level | 0, 3, 6, 12months
  IGF1 level in serum of the enrolled participants

SECONDARY OUTCOMES:
E2 level | 0, 3, 6, 12 months
  serum estrogen level in enrolled participants
LVPWs | 0, 3, 6, 12 months
  left ventricular posterior wall thickness in systolic state
LVIDd | 0, 3, 6, 12 months
  left ventricular internal diameters in diastolic state
LVIDs | 0, 3, 6, 12 months
  left ventricular internal diameters in systolic state
IVSTd | 0, 3, 6, 12 months
  Interventricular septum in diastolic state
IVSTs | 0, 3, 6, 12 months
  Interventricular septum in systolic state
E/e' | 0, 3, 6, 12 months
  the velocity of early diastolic blood flow at the apex of the mitral valve versus the velocity of early diastolic myocardial movement at the annulus of the mitral valve

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong-Shenzhen Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
IPD might not be shared for the candidates' personal privacy